CLINICAL TRIAL: NCT02554240
Title: Active-controlled, Dose-Response, Randomized, Double-blind, Therapeutic Exploratory Clinical Trial to Evaluate the Efficacy and Safety of Intra-articular DA-5202 in Patients With Osteoarthritis of the Knee
Brief Title: Study to Evaluate the Efficacy and Safety of Intra-articular DA-5202 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA5202_KOA_II
Record Dates: First submitted 2015-04-28; First posted 2015-09-18 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- DA-5202 High dose (Experimental): - DA-5202 20mg
  Interventions: Drug: DA-5202 20mg
- DA-5202 Low dose (Experimental): - DA-5202 10mg
  Interventions: Drug: DA-5202 10mg
- Na Hyaluronate 20mg (Active Comparator): Na Hyaluronate 20mg
  Interventions: Drug: Na Hyaluronate 20mg

INTERVENTIONS:
Drug: DA-5202 20mg — once a week, intra-articular injection, for 3 weeks
  Other Names: DA-5202 high dose
  Arms: DA-5202 High dose
Drug: DA-5202 10mg — once a week, intra-articular injection, for 3 weeks
  Other Names: DA-5202 low dose
  Arms: DA-5202 Low dose
Drug: Na Hyaluronate 20mg — once a week, intra-articular injection, for 3 weeks
  Other Names: Hyruan Plus®
  Arms: Na Hyaluronate 20mg

SUMMARY:
This Phase II clinical study is to evaluate the efficacy and safety of DA-5202 in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
Eligible subjects are randomly assigned to receive DA-5202 high dose(20mg) or DA-5202 low dose(10mg) or Na Hyaluronate once a week intra-articular injection for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between 20 and 80 y old
* primary knee osteoarthritis confirmed clinically and radiologically according to American College of Rheumatology criteria and have following 3 items

  1. knee joint pain
  2. have any of the following

     1. males and females more than 50 y
     2. morning stiffness within 30 minutes
     3. crepitus
  3. presence of spur on radiological evidence
* Kellgren-Lawrence Grade Ⅰ to Ⅲ confirmed radiologically
* knee pain under weight-bearing greater than 40/100mm-VAS(Visual Analogue Scale) at randomization visit
* patients willing and able to provide signed informed consent after the nature of the study has been explained

Exclusion Criteria:

* BMI(Body Mass Index) > 32
* complete obliteration of femoropatellar joint space on X-ray
* Kellgren-Lawrence Grade IV
* knee surgery within a year
* history of fracture, rheumatoid arthritis or other inflammatory arthritis in knee articular cavity
* intra-articular corticosteroid injection within 3 months or hyaluronate injection within 6 months
* skin diseases or infection overlying the joint
* history of severe drug allergy or hypersensitivity to drugs(piroxicam, hyaluronic acid)
* history of allergy, asthma, rhinitis, angioedema, rash to aspirin or other NSAIDs (including COX-2 inhibitor)
* treatment with anticoagulants such as heparin or coumarins (warfarin etc.)
* History of GI diseases such as peptic ulcer, bleeding, perforation, ulcerative colitis, Crohn's disease within 1 year
* severe hypertension
* patients with psychiatric disorder, alcoholism, drug addiction
* presence of severe concomitant diseases or malignancy within 5 years
* have participated in another clinical trial 4 weeks prior to the study
* women of child-bearing potential who are not using *adequate means of contraception (*adequate means of contraception: condom, oral contraception, barrier methods using spermicide, intrauterine devices etc.)
* any condition that, in the view of the investigator, would interfere with study participation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2014-12-23 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-10-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline of 100mm-VAS about weight bearing pain in study knee at week 3 | week 3

SECONDARY OUTCOMES:
Change from baseline of 100mm-VAS about Weight bearing pain in study knee at week 1,2,7,12 | week 1,2,7,12
Change from baseline of 100mm-VAS about Resting pain in study knee at week 1,2,3,7,12 | week 1,2,3,7,12
knee joint range of motion change (Observation by investigator) | 24 weeks
knee joint effusion change (Observation by investigator) | 24 weeks
overall assessment of subject and investigator (5-Likert scale) | week 1,2,3,7,12
Change from baseline of 100mm-VAS about Motion pain in study knee at week 1,2,3,7,12 | week 1,2,3,7,12
Change from baseline of 100mm-VAS about Night pain in study knee at week 1,2,3,7,12 | week 1,2,3,7,12
Change from baseline of WOMAC Index total score at Week 1,2,3,7,12 | week 1,2,3,7,12

CONTACTS AND LOCATIONS:
Overall Officials: Myung chul Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea